CLINICAL TRIAL: NCT03809091
Title: Whole Genome Sequencing of Korean Patients With Idiopathic Bronchiectasis for Identification of Disease-Causing Variants
Brief Title: WGS of Korean Idiopathic Bronchiectasis
Acronym: WGS_UNK_BE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: WGS_UNK_BE
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Bronchiectasis Idiopathic; Cystic Fibrosis; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — DNA will be extracted from whole blood samples of patients and their family.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bronchiectasis: The patient with bronchiectasis who has no apparent bronchiectasis-causing etiology will be enrolled. The patient's family who has no bronchiectasis will be also enrolled to identify the patient-specific variants.
  Interventions: Diagnostic Test: Whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Whole genome sequencing — Whole genome sequencing of patients and their family will be performed. Among the variants detected by WGS, disease-causing variants will be analyzed by using segregation analysis.

SUMMARY:
Whole genome sequencing of Korean patients with idiopathic bronchiectasis and their family will perform to identify disease-causing variants.

DETAILED DESCRIPTION:
Idiopathic bronchiectasis may be a manifestation of genetic diseases such as cystic fibrosis, primary ciliary dyskinesia, etc. Diagnosis of these rare genetic diseases is crucial not only because some of the rare diseases developed already effective treatment options, but also the detection of syndrome enables us to detect other organ damages before the deterioration of them.

Several diagnostic tools have been developed; however, the genetic panel has limited screening efficacy due to the genetic heterogeneity of diseases. Even more, especially in Korea, the incidence of idiopathic bronchiectasis caused by the genetic disease is rare, most clinics have limited to assess specialized diagnostic tools such as the specialized genetic panels, sweat chloride test, and the electromagnetic detection tools for ciliary movement.

Whole genome sequencing may be an excellent solution to identify the neglected genetic diseases causing idiopathic bronchiectasis and explore the heterogeneity of disease-causing variants in Korean patients.

ELIGIBILITY:
Inclusion Criteria:

* If the patient has bronchiectasis proved by computed tomography (CT).
* The clinical features of the patient are suitable for ciliary dysfunction disease (primary ciliary dyskinesia, cystic fibrosis), alpha1-antitrypsin deficiency, and primary immune deficiency (hyper-immunoglobulin E syndrome, hypogammaglobulinemia, activated phosphoinositide 3-kinase (PI3K) delta syndrome, bare lymphocyte syndrome)
* The patient has no apparent medical events causing bronchiectasis.

Exclusion Criteria:

* If the patient does not agree or withdraw
* If the patient has any clear etiology causing bronchiectasis including AIDS, malignancy, receiving immunosuppressant or chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients visiting Seoul National Univerisity Hospital outpatient clinic, bronchiectasis patients who have no clear etiology of bronchiectasis and their family will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of diagnosed patients by using whole genome sequencing | 3 years
  The primary objective of this study is to evaluate the effectiveness of whole-genome sequencing (WGS) for idiopathic bronchiectasis patients in Korea. The number of patients newly diagnosed with WGS who are previously not diagnosed will be the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-June Yim, MD, Principal Investigator — Division of Pulmonology and Critical Care Medicine, Seoul National University College of Medicine
Locations (1):
- Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn SJ, Floto AR, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher PW, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society Guideline for bronchiectasis in adults. Thorax. 2019 Jan;74(Suppl 1):1-69. doi: 10.1136/thoraxjnl-2018-212463. No abstract available. PMID 30545985
- [Background] Lonni S, Chalmers JD, Goeminne PC, McDonnell MJ, Dimakou K, De Soyza A, Polverino E, Van de Kerkhove C, Rutherford R, Davison J, Rosales E, Pesci A, Restrepo MI, Torres A, Aliberti S. Etiology of Non-Cystic Fibrosis Bronchiectasis in Adults and Its Correlation to Disease Severity. Ann Am Thorac Soc. 2015 Dec;12(12):1764-70. doi: 10.1513/AnnalsATS.201507-472OC. PMID 26431397
- [Background] Chandrasekaran R, Mac Aogain M, Chalmers JD, Elborn SJ, Chotirmall SH. Geographic variation in the aetiology, epidemiology and microbiology of bronchiectasis. BMC Pulm Med. 2018 May 22;18(1):83. doi: 10.1186/s12890-018-0638-0. PMID 29788932
- [Background] Splinter K, Adams DR, Bacino CA, Bellen HJ, Bernstein JA, Cheatle-Jarvela AM, Eng CM, Esteves C, Gahl WA, Hamid R, Jacob HJ, Kikani B, Koeller DM, Kohane IS, Lee BH, Loscalzo J, Luo X, McCray AT, Metz TO, Mulvihill JJ, Nelson SF, Palmer CGS, Phillips JA 3rd, Pick L, Postlethwait JH, Reuter C, Shashi V, Sweetser DA, Tifft CJ, Walley NM, Wangler MF, Westerfield M, Wheeler MT, Wise AL, Worthey EA, Yamamoto S, Ashley EA; Undiagnosed Diseases Network. Effect of Genetic Diagnosis on Patients with Previously Undiagnosed Disease. N Engl J Med. 2018 Nov 29;379(22):2131-2139. doi: 10.1056/NEJMoa1714458. Epub 2018 Oct 10. PMID 30304647
- See also: Whole genome sequencing enables definitive diagnosis of Cystic Fibrosis and Primary Ciliary Dyskinesia, bioRxiv, 2018 — https://doi.org/10.1101/438838